CLINICAL TRIAL: NCT06335745
Title: A Randomized Phase II Trial Evaluation of the Addition of the Pediatric Cancer Resource Equity (PediCARE) Health Equity Intervention to Usual Supportive Care for Children With Newly Diagnosed High-Risk Neuroblastoma
Brief Title: PediCARE Health Equity Intervention in High-Risk Neuroblastoma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study halted prematurely, prior to enrollment of first participant
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Kira Bona, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-066
Record Dates: First submitted 2024-03-14; First posted 2024-03-28 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Neuroblastoma; High-risk Neuroblastoma; Pediatric Cancer; Disparities; Financial Stress; Poverty
Keywords: Neuroblastoma; High-Risk Neuroblastoma; Disparities; Pediatric cancer; Financial stress; Poverty
MeSH Terms: conditions — Neuroblastoma; Neoplasms; Financial Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: PediCARE + Usual Supportive Care Experimental (Experimental): Participants will be randomized in a 1:1 ratio and stratified according to treatment group and household material hardship (HMH) severity group and participant parents/guardians will complete:
  * Remote baseline visit with introduction to PediCARE intervention by central study team
  * Parent completion of baseline survey.
  * Receipt of monthly PediCARE resource provisions x 6-months.
  * Parent completion of 3-month follow-up survey.
  * Parent completion of 6-month follow up survey and end of intervention period.
  Interventions: Behavioral: PediCARE Intervention
- Arm 2: Usual Supportive Care Arm (No Intervention): Participants will be randomized in a 1:1 ratio and stratified according to treatment group and HMH severity group and participant parent/guardians will complete:
  * Remote baseline visit
  * Parent completion of baseline survey.
  * Receipt of site-specific routine supportive care x6-month study period
  * Parent completion of 3-month follow-up survey
  * Parent completion of 6-month follow-up survey

INTERVENTIONS:
Behavioral: PediCARE Intervention — A household material hardship intervention with monthly, direct provision of groceries and transportation. Resources will be centrally administered by the Dana-Farber Cancer Institute study team.
  Other Names: PediCARE
  Arms: Arm 1: PediCARE + Usual Supportive Care Experimental

SUMMARY:
This is a randomized Phase II trial evaluating the addition of the Pediatric Cancer Resource Equity (PediCARE) health equity intervention to usual supportive care for poverty-exposed children with newly diagnosed high-risk neuroblastoma.

The names of the intervention groups in this research study are:

* Usual supportive care
* PediCARE + usual supportive care

DETAILED DESCRIPTION:
This is a randomized Phase II trial evaluating the addition of the Pediatric Cancer Resource Equity (PediCARE) health equity intervention to usual supportive care for poverty-exposed children with newly diagnosed high-risk neuroblastoma.

Participants will be randomized into one of two groups: Usual Supportive Care vs. PediCARE + Usual Supportive Care. Randomization means a participant is placed into a group by chance.

Participation in this research study is expected to last 6-months.

It is expected about 130 people will participate in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a new diagnosis of high-risk neuroblastoma.
* Patient must be enrolled on APEC14B1 and must have consented to future contact on APEC14B1.
* Patient must be enrolled on ANBL2131.
* Patient aged 0-17 years at the time of consent to ANBL2131.
* Patient must have opted-in to embedded optional ANBL2131 Household Survey.
* Family screened positive for HMH or low-income on ANBL2131 Household Survey. *
* Patient has not yet initiated Induction Cycle 3 on ANBL2131.
* Patient being treated at a U.S. site.
* Patients of all languages are eligible to participate.

  * Eligibility based on Household Survey will be determined by central study team review. HMH exposure will be operationalized as the report of at least one of the following four concrete resource insecurities: (1) Food insecurity, (2) Housing Insecurity, (3) Utility Insecurity, (4) Transportation Insecurity. Low-income will be defined as reported annual household income of less than 200% federal poverty level (FPL).

Exclusion Criteria:

-Patient has transferred to ANBL1531 Arm E.

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2024-09 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Change in Kessler-6 Psychological Distress Scale Score | At baseline and 3 months
  As measured by the Kessler-6 Psychological Distress Scale (K6), a 6-item measure for the level of psychological distress in the past month. Responses are scored on a 5-point Likert scare with answers ranging from 0 "None of the time" to 4 "All of the time," and with a total score range of 0 - 4. Scores > or = 7 suggest "high" distressed and those > or = 13 meet criteria for serious or debilitating psychological distress. A t-test of differences in mean change scores of parent/guardian psychological distress from T1 (baseline) to T2 (3 months) will be used to compare across PediCARE and usual supportive care arms. The distribution of parent psychological distress scores across PediCARE and usual supportive care arms will also be descriptively characterized. The descriptive analyses will be intention-to-treat, defined as all randomized participants with at least one post-baseline contact or follow-up measure.

SECONDARY OUTCOMES:
Proportion of Enrolled Participants (Feasibility) | 5 years
  Feasibility of conducting a centrally-administered companion health equity intervention study among COG trial-enrolled participants will be described using proportions and 95% confidence intervals. Successful feasibility is defined as >75% consent to participation and randomization and <20% attrition. Feasibility metrics will be collected and monitored in real time throughout the duration of the study (about 5 years). An interim analysis for early stopping will also be conducted halfway through accrual (n=40 participants) to assess futility of the feasibility endpoint.
Change in Mean Household Material Hardship (HMH) Score | At baseline and 3-months
  Household Material Hardship (HMH) information will via parent/guardian-completed survey instruments using standardized measures of housing, food, utility, and transportation insecurity. HMH scores will be calculated based on parent/guardian responses and will range from 0-4 based on the number of discrete areas of insecurity endorsed by participants. A t-test of differences in mean HMH change scores from T1 (baseline) to T2 (month 3) will be used to compare across PediCARE and usual supportive care arms. Investigators will also characterize the distribution between T1 and T2 HMH scores across PediCARE and usual supportive care arms on the ordinal scale from 0 to 4 using a chi-square test.

CONTACTS AND LOCATIONS:
Overall Officials: Kira Bona, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to the study PI Dr. Kira Bona. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu